CLINICAL TRIAL: NCT00692042
Title: A Phase I, First Time in Man, Single-Centre, Randomised, Double-Blind (Within Panels), Placebo-Controller Study to Investigate Safety, Tolerability and Pharmacokinetics of AZD1704 After Administration of Oral Single Ascending Doses in Healthy Volunteers
Brief Title: Study to Investigate Safety, Tolerability and Pharmacokinetics of a Single Ascending Dose of AZD1704
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Rolf Karlsten, MD, PhD, Medical Science Director, Emerging Analgesia, Neuroscience, AstraZeneca R&D Södertälje, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: D0980C00001
Record Dates: First submitted 2008-06-05; First posted 2008-06-06 (Estimated); Last update posted 2008-06-24 (Estimated); Status verified 2008-06

CONDITIONS: Pain
Keywords: Safety; tolerability
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AZD1704

INTERVENTIONS:
Drug: AZD1704 — One dose, by mouth

SUMMARY:
The primary aim for this study is to investigate the safety and tolerability of the AZD1704, first time in man.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, man or woman of non child-bearing potential
* Provision of signed informed consent.

Exclusion Criteria:

* History of somatic disease/condition that may interfere with the objectives ot the study, as judged by the Investigator. History of seizures, with the exception of single occasions fever induced seizures in childhood.
* History of previous or ongoing psychiatric disease/condition including psychosis, affective disorder, anxiety disorder, borderline state and personality disorder according to the criteria in the DSM of Mental Disorder, 4th edition
* History of use of antipsychotic, antidepressant or anxiolytic drugs for the treatment of psychiatric disease or symptoms, prescribed as well as non-prescribed use.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2008-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of AZD1704 following single ascending doses in healthy volunteers. | At screening, during residential period (daily) and at follow-up

SECONDARY OUTCOMES:
To investigate the subjective CNS effects of specific adjectives (stimulated, anxious, sedated, down and high) rated on visual analogue mood scale (VAMS). | During residential period (daily)

CONTACTS AND LOCATIONS:
Overall Officials: Billy Fahy, MD, Principal Investigator — AstraZeneca R&D CPU Nottingham, UK; Lars Ståhle, MD, Study Chair — AstraZeneca R&D Södertälje, Sweden
Locations (1):
- Reserach Site, Macclesfield, Cheshire, United Kingdom